CLINICAL TRIAL: NCT06508268
Title: Language, Speech and Motor Function in Mild Cognitive Impairment Due to AD and Alzheimer's Disease
Brief Title: Language, Speech and Motor Function in MCI Due to AD and Alzheimer's Disease
Status: Recruiting | Type: Observational
Sponsor: Hanze University of Applied Sciences Groningen (Other)
Collaborators: University of Groningen (Other)
Responsible Party: Principal Investigator, Hans Hobbelen, Professor, Hanze University of Applied Sciences Groningen
Other Study IDs: NL79836.042.23
Record Dates: First submitted 2024-05-22; First posted 2024-07-18 (Actual); Last update posted 2024-07-18 (Actual); Status verified 2024-07

CONDITIONS: Alzheimer's Disease; MCI Due to AD; Dementia Alzheimers
Keywords: Alzheimer's disease; MCI due to AD; Language; Speech; Motor; Gait; Hand grip strength; Fluency
MeSH Terms: conditions — Alzheimer Disease; Language; Speech

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Persons with Mild Cognitive Impairment due to AD
  Interventions: Behavioral: GAITRite walkway system OR 4-meter walking speed test; Behavioral: Jamar hand dynamometer; Behavioral: Picture description task; Behavioral: Autobiographical semi-structured conversation; Behavioral: Verbal fluency
- Persons with mild AD
  Interventions: Behavioral: GAITRite walkway system OR 4-meter walking speed test; Behavioral: Jamar hand dynamometer; Behavioral: Picture description task; Behavioral: Autobiographical semi-structured conversation; Behavioral: Verbal fluency
- Persons with moderate AD
  Interventions: Behavioral: GAITRite walkway system OR 4-meter walking speed test; Behavioral: Jamar hand dynamometer; Behavioral: Picture description task; Behavioral: Autobiographical semi-structured conversation; Behavioral: Verbal fluency
- Persons without cognitive impairment, age-matched with persons with MCI due to AD and AD
  Interventions: Behavioral: GAITRite walkway system OR 4-meter walking speed test; Behavioral: Jamar hand dynamometer; Behavioral: Picture description task; Behavioral: Autobiographical semi-structured conversation; Behavioral: Verbal fluency

INTERVENTIONS:
Behavioral: GAITRite walkway system OR 4-meter walking speed test — Gait will be assessed by the GAITRite walkway system OR the 4-meter walking speed test
Behavioral: Jamar hand dynamometer — Hand grip strength will be assessed by a Jamar hand dynamometer
Behavioral: Picture description task — Characteristics Dutch/Frisian language Language and speech will be assessed by the Cookie Theft Picture-task (a picture description task from Berube et al., 2019)
  Other Names: Cookie Theft Picture
Behavioral: Autobiographical semi-structured conversation — Characteristics Dutch/Frisian language and speech will be assessed by an autobiographical semi-structured conversation
Behavioral: Verbal fluency — The mental lexicon of Dutch/Frisian language will be assessed by a two verbal fluency tests, including letter fluency and categorical fluency

SUMMARY:
The goal of this observational cross-sectional study is to explore the characteristics of language, speech, and motor function in persons with Mild Cognitive Impairment due to Alzheimer's disease ("MCI due to AD") and persons with mild and moderate Alzheimer's disease ("AD"). This study aims to:

* Explore motor, speech, and language functions in MCI due to AD and mild and moderate AD.
* Combine the characteristics of motor, language, and speech functions to gain more insight into the association of language, speech, and motor changes during MCI due to AD and mild and moderate AD.

Researchers will compare the outcomes to an age-matched control group without cognitive impairment.

Participants will undergo:

* Two motor function tests to assess gait and hand grip strength.
* Four language and speech function tests to assess spontaneous speech and verbal fluency..

ELIGIBILITY:
Inclusion Criteria:

A subject with MCI with a likelihood of underlying AD pathophysiology must meet the following criteria:

* Established diagnosis of MCI due to AD with a likelihood according to NIA-AA criteria (Albert et al., 2011).
* A score of stage three on the Global Deterioration Scale (GDS) (Reisberg et al., 1982).

A subject with AD must meet the following criteria:

* Established diagnosis of AD (amnestic or non-amnestic) or etiologically mixed presentation of AD according to DSM-5 (American Psychiatric Association, 2013) or NINCDS-ARDRA criteria (Jack et al., 2018; McKann et al., 2011).
* The following scores on the Global Deterioration Scale (GDS): four for mild AD, five for moderate AD (Reisberg et al., 1982).

All subjects of the control group must meet the following criteria:

* A score of stage one or two on the Global Deterioration Scale (GDS) (Reisberg et al., 1982).
* They are age-matched with the MCI due to AD or AD patients included in the study.

All subjects must meet the following criteria:

* First language is Dutch and/or Frisian.
* Able to walk independently with or without walking aid.
* Able to squeeze with each hand.

Exclusion Criteria:

A subject with MCI due to AD or AD who meets the following criteria will be excluded from participation in this study:

* Having a neurological or neurodegenerative disease or disorder that may be contributing to cognitive impairment above and beyond that caused by AD or mixed AD; Down's syndrome, other subtypes of dementia, autism spectrum disorder.
* Having an established diagnosis of a psychiatric disorder, e.g. schizophrenia, depression.

All subjects in the control group who meets following criteria will be excluded from participation in this study:

● Suffers from a neurological, neurodegenerative or psychiatric disease or disorder.

All subjects in any group who meet any of the following criteria will be excluded from participation in this study:

* Hearing loss (with or without hearing aid) that affects communication.
* Vision loss (with or without glasses or lenses) that affects communication.
* History of language problems, speech problems or dyslexia.
* Suffers from additional disorders or diseases which may limit gait, hand grip strength, language and/or speech.
* Medication use that influence gait, hand grip strength, speech or language performance at time of testing.
* Being terminally ill (i.e., life expectancy < 2 weeks according to the attending physician).

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The envisaged total participants of this study is: 52 persons with MCI due to AD, 52 persons with mild AD, 52 persons with moderate AD, 52 and 52 age-matched persons without cognitive impairment. The first language of the participants is either Frisian and/or Dutch. The participants may in addition to that also speak a Dutch dialect or another language
Sampling Method: Non-Probability Sample
Enrollment: 208 (Estimated)
Dates: Start 2024-07-12 (Estimated); Primary Completion 2025-02-09 (Estimated); Study Completion 2025-02-09 (Estimated)

PRIMARY OUTCOMES:
Language and speech characteristics of spontaneous speech | 4 months
  Autobiographical semi-structured interview and a picture description task ("The Cookie Theft Picture (Berube et al., 2019))
Verbal fluency | 4 months
  Naming animals and professions
Letter fluency | 4 months
  Naming letters starting with the letters D and A
Temporal and spatial parameters of gait | 4 months
  Gaitrite walkway system (GAITRite) or 4-meter walking speed test
Hand grip strength | 4 months
  Jamar hand dynamometer

CONTACTS AND LOCATIONS:
Locations (1):
- Hanze University, Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided
This study is based on FAIR principles (Findable, Accessible, Interoperable and Reusable). This means that, all anonymized data and meta-data will be archived and shared during or after 5 years after completion of this study in one or more of the following database systems: Faith Research (https://www.faithresearch.nl/), DANS ('Data Archiving and Networked Services) and DataverseNL (https://dataverse.nl).